CLINICAL TRIAL: NCT05414110
Title: Effect of Airway Pressure Release Ventilation(APRV) on Right Ventricular Function Assessed by Transthoracic Echocardiography
Brief Title: Effect of Airway Pressure Release Ventilation on Right Ventricular Function Assessed by Transthoracic Echocardiography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: TTEC20220103
Record Dates: First submitted 2022-04-05; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Ventilation Therapy; Complications; Right Ventricular Function; ARDS; Transthoracic Echocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Effects of APRV on right ventricular function in patients with acute respiratory distress syndrome by transthoracic echocardiography

DETAILED DESCRIPTION:
Effects of APRV on right ventricular function in patients with acute respiratory distress syndrome(ARDS) by transthoracic echocardiography，which includes TAPSE, S' by TDI, RV FAC, tricuspid regurgitation,RVEDA/LVEDA,RV, Velocity time integration(VTI) of the left ventricular outflow tract blood flow.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the 2012 Berlin ARDS diagnostic criteria and undergo invasive mechanical ventilation
2. PEEP≥5cmH2O, oxygenation index≤200mmHg
3. Endotracheal intubation and mechanical ventilation time <48h
4. Age ≥18 years old and ≤80 years old

Exclusion Criteria:

1. Aged less than 18 years old or older than 80 years old
2. Obese patients with BMI≥35kg/m2;
3. Pregnant and lactating women
4. The expected time of invasive mechanical ventilation is expected to be less than 48h
5. Neuromuscular disease known to require prolonged mechanical ventilation
6. Severe chronic obstructive pulmonary disease
7. Intracranial hypertension
8. Bullae or pneumothorax, subcutaneous emphysema, mediastinal emphysema
9. extracorporeal membrane oxygenation(ECMO) has been performed when entering the ICU
10. Refractory shock
11. Severe cardiac dysfunction (New York Heart Association class III or IV, acute coronary syndrome or persistent ventricular tachyarrhythmia), right heart enlargement due to chronic cardiopulmonary disease, cardiogenic shock or heart enlargement postoperative;
12. Failure to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Include as many eligible study populations as possible by study protocol
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-03 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Right ventricular area fractional change (RV FAC) | RV FAC monitoring was performed 1 day after APRV mechanical ventilation
  Right ventricular area fractional change (RV FAC)is a simple and repeatable ultrasound method for evaluating RV function. Methods: The RV end-diastolic area (RVEDA) and RV end-systolic area (RVESA) were measured on the apical four-chamber section by two-dimensional ultrasound. RV FAC=(RVEDA- RVESA)/RVEDA*100%.
Tricuspid annular systolic displacement(TAPSE) | TAPSE monitoring was performed 1 day after APRV mechanical ventilation
  TAPSE:TAPSE is one of the most effective ultrasound methods for evaluating right ventricular function.Measurement method: TAPSE was measured on the four-chamber section of the apex of the heart by M-mode ultrasound. the sampling line was placed at the side wall of the tricuspid valve ring, parallel to the free wall of the right ventricle as far as possible, and the displacement of the tricuspid valve ring was measured from the end of diastole to the end of systole.
Tricuspid annular systolic S' velocity (TS') | TS' monitoring was performed 1 day after APRV mechanical ventilation
  TS' is an objective and accurate ultrasound technique for evaluating right ventricular function.Measurement method:The sample volume was applied to the free wall of the RV and the peak velocity of tricuspid annulus motion was measured in the four-chamber section of the apex by tissue doppler imaging (TDI).
Right ventricular end-diastolic area/left ventricular end-diastolic area (RVEDA/LVEDA) | RVEDA/LVEDA monitoring was performed 1 day after APRV mechanical ventilation
  RVEDA/LVEDA a simple and repeatable ultrasound method for evaluating dynamics changes of RV function.Methods: The RV end-diastolic area (RVEDA) and left ventricular(LV) end-systolic area (LVEDA) were measured on the apical four-chamber section by two-dimensional ultrasound.
Pulmonary circulatory resistance (PVR) | PVR monitoring was performed 1 day after APRV mechanical ventilation
  Increased PVR can lead to deterioration of RV function.Pulse Doppler imaging (PWD) was used to obtain the pulmonary artery flow spectrum from the pulmonic valve on the short axial section of the parasternal great vessels.

SECONDARY OUTCOMES:
Heart rate (HR) | HR monitoring was performed before APRV mechanical ventilation and 6 hours, 12 hours, Day 1, Day 2, Day 3 after APRV mechanical ventilation, and 24 hours after APRV ended
  HR is a basic element of hemodynamic index
Systolic blood pressure (SBP) | SBP monitoring was performed before APRV mechanical ventilation and 6 hours, 12 hours, Day 1, Day 2, Day 3 after APRV mechanical ventilation, and 24 hours after APRV ended
  SBP is basic element of hemodynamic index
Mean arterial pressure (MAP) | MAP monitoring was performed before APRV mechanical ventilation and 6 hours, 12 hours, Day 1, Day 2, Day 3 after APRV mechanical ventilation, and 24 hours after APRV ended
  MAP represents peripheral organ perfusion pressure
cardiac output (CO) | CO monitoring was performed before APRV mechanical ventilation and 6 hours, 12 hours, Day 1, Day 2, Day 3 after APRV mechanical ventilation, and 24 hours after APRV ended by ultrasound
  CO is an important parameter to reflect the cardiac function of patients
Stroke volume (SV) | SV monitoring was performed before APRV mechanical ventilation and 6 hours, 12 hours, Day 1, Day 2, Day 3 after APRV mechanical ventilation, and 24 hours after APRV ended by ultrasound
  Stroke volume is the amount of blood that the ventricle shoots out during a single heart beat.
28-day mortality | Day 28 after study entry
  28-day mortality after study entry
The number of days in ICU | From the day subjects entered ICU to the day left ICU(up to 90 days)
  The number of days in ICU(up to 90 days)
The number of days in hospital | From the day subjects entered hospital to the day left hospital including death(up to 90 days)
  The number of days in hospital(up to 90 days)
in-hospital mortality | From the day patients admitted to hospital to the day death or discharge(up to 90 days)
  Any death occurred during hospitalization(up to 90 days)
Sequential Organ Failure Assessment score | Within 2 hours admission to ICU and 24 hours after inclusion in the study
  The higher the Sequential Organ Failure Assessment(SOFA) score, the higher the disease risk factor and the higher the mortality rate(The highest score is 24, while the lowest score is 0).
Acute Physiology and Chronic Health Evaluation II score | Within 2 hours admission to ICU and 24 hours after inclusion in the study
  The higher the Acute Physiology and Chronic Health Evaluation II(APACHE II) score, the higher the disease risk factor and the higher the mortality rate(the highest score is 71, while the lowest score is 0).In particular, the accuracy of group patient prediction is high.
the effect of APRV ventilation time on right ventricular area fractional change (RV FAC) in ARDS patients | RV FAC monitoring was performed before APRV mechanical ventilation and 6 hours, 12 hours, Day 1, Day 2, Day 3 after APRV mechanical ventilation, and 24 hours after APRV ended by ultrasound
  The RV end-diastolic area (RVEDA) and RV end- systolic area (RVESA) were measured on the apical four-chamber section by two-dimensional ultrasound. RV FAC=(RVEDA- RVESA)/RVEDA*100%.
the effect of APRV ventilation time on tricuspid annular systolic displacement (TAPSE) in ARDS patients. | TAPSE monitoring was performed before APRV mechanical ventilation and 6 hours, 12 hours, Day 1, Day 2, Day 3 after APRV mechanical ventilation, and 24 hours after APRV ended by ultrasound
  TAPSE was measured on the four-chamber section of the apex of the heart by M-mode ultrasound. the sampling line was placed at the side wall of the tricuspid valve ring, parallel to the free wall of the right ventricle as far as possible, and the displacement of the tricuspid valve ring was measured from the end of diastole to the end of RV systole.
the effect of APRV ventilation time on tricuspid annular systolic S' velocity in ARDS patients. | Tricuspid annular systolic S' velocity monitoring was performed before APRV mechanical ventilation and 6 hours, 12 hours, Day 1, Day 2, Day 3 after APRV mechanical ventilation, and 24 hours after APRV ended by ultrasound
  Tricuspid annular systolic S' velocity is an objective and accurate ultrasound technique for evaluating right ventricular function.Measurement method:The sample volume was applied to the free wall of the RV and the peak velocity of tricuspid annulus motion was measured in the four-chamber section of the apex by tissue doppler imaging (TDI).
the effect of APRV ventilation time on right ventricular end-diastolic area/left ventricular end-diastolic area (RVEDA/LVEDA) in ARDS patients. | RVEDA/LVEDA monitoring was performed before APRV mechanical ventilation and 6 hours, 12 hours, Day 1, Day 2, Day 3 after APRV mechanical ventilation, and 24 hours after APRV ended by ultrasound
  RVEDA/LVEDA：RVEDA/LVEDA a simple and repeatable ultrasound method for evaluating dynamics changes of RV function.Methods: The RV end-diastolic area (RVEDA) and LV end-systolic area (lVEDA) were measured on the apical four-chamber section by two-dimensional ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: xiaojing zou, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang H, Huang W, Zhang Q, Chen X, Wang X, Liu D; Critical Care Ultrasound Study Group. Prevalence and prognostic value of various types of right ventricular dysfunction in mechanically ventilated septic patients. Ann Intensive Care. 2021 Jul 13;11(1):108. doi: 10.1186/s13613-021-00902-9. PMID 34255224
- [Result] Boissier F, Katsahian S, Razazi K, Thille AW, Roche-Campo F, Leon R, Vivier E, Brochard L, Vieillard-Baron A, Brun-Buisson C, Mekontso Dessap A. Prevalence and prognosis of cor pulmonale during protective ventilation for acute respiratory distress syndrome. Intensive Care Med. 2013 Oct;39(10):1725-33. doi: 10.1007/s00134-013-2941-9. Epub 2013 May 15. PMID 23673401
- [Result] Dong D, Zong Y, Li Z, Wang Y, Jing C. Mortality of right ventricular dysfunction in patients with acute respiratory distress syndrome subjected to lung protective ventilation: A systematic review and meta-analysis. Heart Lung. 2021 Sep-Oct;50(5):730-735. doi: 10.1016/j.hrtlng.2021.04.011. Epub 2021 Jun 9. PMID 34118786
- [Result] Mekontso Dessap A, Boissier F, Charron C, Begot E, Repesse X, Legras A, Brun-Buisson C, Vignon P, Vieillard-Baron A. Acute cor pulmonale during protective ventilation for acute respiratory distress syndrome: prevalence, predictors, and clinical impact. Intensive Care Med. 2016 May;42(5):862-870. doi: 10.1007/s00134-015-4141-2. Epub 2015 Dec 9. PMID 26650055
- [Result] Jardin F, Vieillard-Baron A. Right ventricular function and positive pressure ventilation in clinical practice: from hemodynamic subsets to respirator settings. Intensive Care Med. 2003 Sep;29(9):1426-34. doi: 10.1007/s00134-003-1873-1. Epub 2003 Aug 9. No abstract available. PMID 12910335
- [Result] Sun X, Liu Y, Li N, You D, Zhao Y. The safety and efficacy of airway pressure release ventilation in acute respiratory distress syndrome patients: A PRISMA-compliant systematic review and meta-analysis. Medicine (Baltimore). 2020 Jan;99(1):e18586. doi: 10.1097/MD.0000000000018586. PMID 31895807
- [Result] Zhou Y, Jin X, Lv Y, Wang P, Yang Y, Liang G, Wang B, Kang Y. Early application of airway pressure release ventilation may reduce the duration of mechanical ventilation in acute respiratory distress syndrome. Intensive Care Med. 2017 Nov;43(11):1648-1659. doi: 10.1007/s00134-017-4912-z. Epub 2017 Sep 22. PMID 28936695

DOCUMENTS (1):
  • Study Protocol (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT05414110/Prot_000.pdf